CLINICAL TRIAL: NCT01809119
Title: Prospective Randomized Study Comparing Laparoscopic Versus Open Partial Nephrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Marcos Francisco Dall'Oglio, M.D. Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UROUSP - 005
Record Dates: First submitted 2013-03-08; First posted 2013-03-12 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Kidney Neoplasms
Keywords: Kidney Neoplasms, Minimally invasive surgery, Renal cell carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic Partial Nephrectomy (Experimental): Patients with kidney neoplasms submitted to laparoscopic partial nephrectomy
  Interventions: Procedure: Partial nephrectomy
- Open Partial Nephrectomy (Active Comparator): Patients with kidney neoplasms submitted to open partial nephrectomy
  Interventions: Procedure: Partial nephrectomy

INTERVENTIONS:
Procedure: Partial nephrectomy

SUMMARY:
Partial nephrectomy is considered the standard treatment for renal tumors smaller than 7 cm. With the evolution of image diagnostic tools and dissemination of its use, smaller tumors are being commonly diagnosed and treated. The partial open nephrectomy is still considered the gold standard technique for nephron sparing surgery, especially when the surgeon is not experienced with the minimally invasive surgery. In the last 15 years, uncountable minimally invasive techniques were developed, including the laparoscopic partial nephrectomy. The objective of this study is compare the partial laparoscopic nephrectomy to open partial nephrectomy in terms of perioperative, oncologic and functional outcomes. A balanced randomized prospective trial will be conducted. One group of patients will be submitted to to open partial nephrectomy while the other group of patients will be submitted to laparoscopic partial nephrectomy. A randomized prospective trial comparing the two techniques is necessary to determine the differences in outcomes between them and if the laparoscopic partial nephrectomy can be performed without harms to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with renal tumor cT1N0M0; (<7 cm)
* Normal renal function (serum creatinine <1.2 and glomerular filtration rate> 60mL/min/1.73m2)
* Tumor only

Exclusion Criteria:

* Functional or anatomical solitary kidney
* Horseshoe kidney, ectopic or malformed
* Clinical contraindication to surgery
* Contraindication to laparoscopic surgery
* Association with other renal pathologies
* Evidence of lymph node or systemic disease in preoperative staging

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2012-12; Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Surgical Complications | 6 months

SECONDARY OUTCOMES:
Renal Function | 2 years
Oncological outcomes | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Marcos F Dall'Oglio, M.D., Associate Professor, Study Director — Cancer Institute of the State of São Paulo - University of Sao Paulo; Giuliano B Guglielmetti, Doctor, Principal Investigator — Cancer Institute of the State of São Paulo - University of Sao Paulo; Alexandre C Sant'Anna, Doctor, Study Chair — Cancer Institute of the State of São Paulo - University of Sao Paulo
Locations (1):
- Cancer Institute of the State of São Paulo, São Paulo, Brazil